CLINICAL TRIAL: NCT05185934
Title: The Effect of Dietary Glycocalyx Precursor Supplementation on Endothelial Function, on Markers of Vascular Function and on Cardiac Performance in Patients With COVID-19 Infection.
Brief Title: The Effect of Dietary Intervation on Endothelial Glycocalyx in COVID-19 Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 668/30-11-2021
Record Dates: First submitted 2022-01-09; First posted 2022-01-11 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Endothelial Dysfunction
Keywords: COVID-19; Arterial Stiffness; Endothelial Glycocalyx; Coronary microcirculation; Left ventricular myocardial deformation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Sixty patients with COVID-19 infection will be randomized to receive food supplement Endocalyx (n=30) or placebo (n=30) for 4 consecutive months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement Endocalyx (Active Comparator): Thirty patients with COVID-19 infection will randomized to receive 4 capsules a day of the food supplement Endocalyx for 4 months.
  Interventions: Dietary Supplement: Food supplement Endocalyx
- Placebo (Placebo Comparator): Thirty patients with COVID-19 infection will randomized to receive 4 capsules a day of the placebo for 4 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement Endocalyx — Patients with COVID-19 infection will be randomized to receive food supplement Endocalyx for 4 months.
  Arms: Food supplement Endocalyx
Dietary Supplement: Placebo — Patients with COVID-19 infection will be randomized to receive placebo for 4 months.
  Arms: Placebo

SUMMARY:
The food supplement Endocalyx is considered to support the endothelial glycocalyx integrity by supplying sulfated polysaccharides, anti-oxidant enzymes and additional substrates for glycocalyx synthesis. The investigators will study the effect of Endocalyx on endothelial, vascular and left ventricular myocardial function in patients with COVID-19 infection.

DETAILED DESCRIPTION:
Sixty patients who have been hospitalized due to COVID-19 infection will be randomized to receive food supplement Endocalyx (4 capsules per day) (n=30) or placebo (n=30) for 4 consecutive months.

ELIGIBILITY:
Inclusion Criteria:

* caucasian patients
* hospitalization for COVID-19 infection
* diagnosis of COVID-19 proven by PCR

Exclusion Criteria:

* Pregnancy and breastfeeding
* Foreseen inability to attend scheduled visits
* History of acute coronary syndrome. Coronary artery disease will be excluded by a clinical history, examination and electrocardiogram.
* Moderate or severe valve disease
* Primary cardiomyopathies
* Chronic obstructive pulmonary disease
* Asthma
* Chronic kidney disease (estimated glomerular filtration rate [eGFR] ≤60 ml/min/1.73 m2)
* Liver failure
* Malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Endocalyx effects on endothelial glycocalyx thickness | four months
  Endocalyx effects on endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels using Sidestream Dark Field (SDF) imaging

SECONDARY OUTCOMES:
Endocalyx effects on arterial stiffness | four months
  Endocalyx effects on arterial stiffness as assessed by carotid to femoral pulse wave velocity (PWV, m/s) using tonometry.
Endocalyx effects on coronary microcirculation | four months
  Endocalyx effects on coronary function as assessed by measuring coronary flow reserve of left anterior descending artery. Coronary flow reserve is estimated by Doppler echocardiography as the ratio of coronary flow velocity (m/s) after bolus intravenous adenosine infusion to coronary flow velocity (m/s) at rest.
Endocalyx effects on left ventricular myocardial function | four months
  Endocalyx effects on left ventricular function as assessed by global longitudinal strain using speckle-tracking echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavlidis G, Kountouri A, Katogiannis K, Thymis J, Nikolaou PE, Chania C, Karalis J, Kostelli G, Michalopoulou E, Katsanaki E, Parissis J, Vink H, Long R, Tsiodras S, Lambadiari V, Ikonomidis I. Effects of 4-month treatment with glycocalyx dietary supplement on endothelial glycocalyx and vascular function after COVID-19 infection. Eur J Clin Invest. 2025 Jul;55(7):e70058. doi: 10.1111/eci.70058. Epub 2025 Apr 24. PMID 40270280